CLINICAL TRIAL: NCT07216989
Title: Fastomics: Metabolic and Therapeutic Effects of Prolonged Fasting
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: MED-2025-33589
Record Dates: First submitted 2025-09-22; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Insulin Resistance; Fasting
MeSH Terms: conditions — Insulin Resistance; Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples will be stored, with participant consent, deidentified in freezers under the care of the PI indefinitely
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 60 Hour Fasting: healthy participants who agree to fast with water for up to 60 hours while wearing continuous glucose monitors
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Fasting — fast with water for up to 60 hours while wearing continuous glucose monitors

SUMMARY:
This is an observational study investigating how the metabolic and cell marker changes in Prolonged Fasting in the serum may be used against a cell-based model of disease for therapeutic purposes.

DETAILED DESCRIPTION:
There is potential benefit to prolonged water fasting, fasting with ad libitum water intake and consciously eating little to no food or caloric beverages, with regards to reducing weight, fat mass, insulin resistance and oxidative stress while improving glycemic control. Multiple studies have shown that prolonged water-only Fasting for 5-20 days has been safe in humans. A minimum of 2-3 liters of water intake daily is recommended by previous studies in which longer periods of up to 8 days fasting were observed. Prolonged fasting (36 hours) in humans upregulated multiple bioactive metabolites in the serum; exposure to this serum extended the lifespan of yeast (Caenorhabditis elegans) by 96%. In patients receiving chemotherapy, extended fasting periods of up to 60 hours (36 hours before and 24 hours after chemotherapy) are well-tolerated and reduce chemotherapy-related side effects, similar to shorter fasting durations of 28-48 hours. Herein, we propose an in-depth evaluation of Prolonged Fasting on serum metabolite measures and the effects of these serum metabolites on different cell-based models of disease (i.e. cancer, metabolic syndrome, diabetes). We hypothesize that Prolonged Fasting will alter serum metabolites to favorably improve cell-based models of disease. The significance of this study is to understand the extent of immune system activation and metabolic changes resulting from Prolonged Fasting. This sets the stage for developing tailored interventions to capture the fasting phenotype without the process of actually fasting.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18-65 years old
* Not pregnant
* No comorbid conditions
* BMI of 18.5-29.9.
* Has a smartphone

Exclusion Criteria:

* Concern for active eating disorder per screening questionnaire
* Self-reported eating disorder or history of eating disorder
* History of hypoglycemia or contraindication for Prolonged Fasting
* Weight <120lbs
* History of blood donation within the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Self-reportedly healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of doing prolonged fasting in this population | Day 4
  measured by % participants completing all the visits

SECONDARY OUTCOMES:
Exposure of plasma on in vitro breast cancer cell models with regards to cell viability, signaling, function, plasma metabolites, and inflammatory markers | Baseline
  Exposure of cancer cell lines in combination with various doses of chemotherapy agents (e.g., doxorubicin). potential example measures include the following: Serum samples will be analyzed with a Meso Scale Discovery V-PLEX Proinflammatory Panel, which measures the following markers of inflammation: IFN-γ, IL-1β, IL- 2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13,TNF-α.
Exposure of plasma on in vitro breast cancer cell models with regards to cell viability, signaling, function, plasma metabolites, and inflammatory markers | After 60 hours of fasting
  Exposure of cancer cell lines in combination with various doses of chemotherapy agents (e.g., doxorubicin). potential example measures include the following: Serum samples will be analyzed with a Meso Scale Discovery V-PLEX Proinflammatory Panel, which measures the following markers of inflammation: IFN-γ, IL-1β, IL- 2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13,TNF-α.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Chow, MD, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States